CLINICAL TRIAL: NCT04128683
Title: Toward Understanding Dopamine Receptor Contributions to Prediction Error and Reversal Learning in Anorexia Nervosa
Brief Title: Dopamine Receptor Contributions to Prediction Error and Reversal Learning in Anorexia Nervosa
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 191348; 5R21MH120475 (NIH)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Amisulpride; Bromocriptine

STUDY DESIGN:
Intervention Model Description: There are two groups in this study, healthy controls and anorexia nervosa. Each group completes 3 MRI scans where one of the following medications are administered 3 hours prior to the start of the scan: placebo, amisulpride, bromocriptine. The order of the medication scans was randomized.
Who Masked: Participant
Masking Description: The participant did not know what medication they were receiving on each scan day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Healthy Controls, Scan1: Placebo; Scan2: Amisulpride; Scan3: Bromocriptine (Experimental): Individuals in the healthy control group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Placebo(single dose, 3 hours pre-scan) Scan 2: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 3: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Healthy Controls, Scan1: Placebo; Scan2: Bromocriptine; Scan3: Amisulpride; (Experimental): Individuals in the healthy control group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Placebo(single dose, 3 hours pre-scan) Scan 2: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 3: Amisulpride (single dose, 400 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Healthy Controls, Scan1: Amisulpride; Scan2: Placebo; Scan3: Bromocriptine (Experimental): Individuals in the healthy control group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 2: Placebo(single dose, 3 hours pre-scan) Scan 3: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Healthy Controls, Scan1: Amisulpride; Scan2: Bromocriptine; Scan1: Placebo (Experimental): Individuals in the healthy control group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 2: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 3: Placebo(single dose, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Healthy Controls, Scan1: Bromocriptine; Scan2: Placebo; Scan 3: Amisulpride (Experimental): Individuals in the healthy control group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 2: Placebo(single dose, 3 hours pre-scan) Scan 3: Amisulpride (single dose, 400 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Healthy Controls, Scan1: Bromocriptine; Scan2: Amisulpride; Scan3: Placebo (Experimental): Individuals in the healthy control group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 2: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 3: Placebo(single dose, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Anorexia Nervosa, Scan1: Placebo; Scan2: Amisulpride; Scan3: Bromocriptine (Experimental): Individuals in the anorexia nervosa group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Placebo(single dose, 3 hours pre-scan) Scan 2: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 3: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Anorexia Nervosa, Scan1: Placebo; Scan2: Bromocriptine; Scan3: Amisulpride; (Experimental): Individuals in the anorexia nervosa group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Placebo(single dose, 3 hours pre-scan) Scan 2: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 3: Amisulpride (single dose, 400 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Anorexia Nervosa, Scan1: Amisulpride; Scan2: Placebo; Scan3: Bromocriptine (Experimental): Individuals in the anorexia nervosa group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 2: Placebo(single dose, 3 hours pre-scan) Scan 3: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Anorexia Nervosa, Scan1: Amisulpride; Scan2: Bromocriptine; Scan1: Placebo (Experimental): Individuals in the anorexia nervosa group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 2: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 3: Placebo(single dose, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Anorexia Nervosa, Scan1: Bromocriptine; Scan2: Placebo; Scan 3: Amisulpride (Experimental): Individuals in the anorexia nervosa group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 2: Placebo(single dose, 3 hours pre-scan) Scan 3: Amisulpride (single dose, 400 mg, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo
- Anorexia Nervosa, Scan1: Bromocriptine; Scan2: Amisulpride; Scan3: Placebo (Experimental): Individuals in the anorexia nervosa group were randomized to the following scan order. Participants were administered a study medication or placebo 3 hours prior to the start of the scan. The participant did not know what study medication they received for each scan:
  Scan 1: Bromocriptine (single dose, 1.25 mg, 3 hours pre-scan) Scan 2: Amisulpride (single dose, 400 mg, 3 hours pre-scan) Scan 3: Placebo(single dose, 3 hours pre-scan)
  Interventions: Drug: amisulpride; Drug: bromocriptine; Drug: Placebo

INTERVENTIONS:
Drug: amisulpride — Dopamine D2 antagonist to test how it affects brain response and behavior to prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
  Other Names: Solian
Drug: bromocriptine — Dopamine D2 receptor agonist test how it affects brain response and behavior to prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
  Other Names: Parlodel
Drug: Placebo — Placebo pill with no active drug ingredients

SUMMARY:
Anorexia nervosa (AN) is an eating disorder associated with intense fear of weight gain, food refusal, and severe weight loss. AN has the highest mortality rate among the psychiatric disorders; however, little is known about biomarkers, and no medication has been approved for AN. Many individuals only partially recover, and treatment options, especially for the psychological components of the illness, are not very effective, highlighting the need for more effective treatments.

Brain reward pathways have a direct impact on the drive to eat, and a variety of neuroimaging studies have suggested altered reward processing in AN. The neurotransmitter dopamine has a central role in the reward circuitry to drive food approach, and the dynamic interplay between dopamine receptor response and food restriction could have implications for the pathophysiology of AN. Dopamine-related brain function has been studied indirectly using functional magnetic resonance brain imaging (fMRI) and tasks that deliver reward stimuli unexpectedly, that elicit the so-called prediction error (PE) response.

Research in AN showed repeatedly altered PE processing suggesting altered dopamine circuit function in the disorder.

Dopamine and PE response have also been associated with altered reversal learning, which has important treatment implication for AN as reversal learning is impaired in the disorder and modulation of the dopamine system could improve treatment.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls

* Females ages 18-29 years
* Healthy body weight between 90 and 110 % average body weight since puberty.
* Regular monthly menstrual cycle
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* English is primary language spoken

Restricting Type Anorexia Nervosa

* Females ages 18-29 years
* Diagnostic criteria. Current diagnosis of AN, including being underweight below 17.5 body mass index (BMI, kg/m2), will have a severe fear of weight gain, body image distortion and absence of the menstrual cycle over three consecutive months.
* First 1-2 weeks in treatment at The University of California San Diego Eating Disorders Center for Treatment and Research or Rady Children's Hospital San Diego Medical Behavioral Unit.
* Restricting subtype, that is without binge/purge behaviors
* Edinburgh Handedness Inventory Revised (EHI-R) LQ* score > +200
* English is primary language spoken

Exclusion Criteria:

Healthy Controls

* Current pregnancy or breast feeding within last 3 months
* Illiterate/Blind individuals
* First degree relative with current or past eating disorder
* Current Medications other than BCP or IUD
* Contraindications to amisulpride or bromocriptine (as determined through medical history in bioscreen and PI interview) including: Syncopal migraine; Uncontrolled hypertension; Pheochromocytoma; Prolactinoma; Breast cancer; hypersensitivity/allergy to amisulpride or bromocriptine; History of long QT syndrome; Family history of sudden death or long QT syndrome; History of seizures or seizure disorder
* Past or present Axis I psychiatric disorder including substance or alcohol use disorder as determined through SCID-5 clinical interview
* Major Medical illness (as determined through medical history in bioscreen and PI interview) such as:

  o Conditions that are life threatening: cancer heart disease stroke HIV/AIDS

  o Conditions that are life threatening Conditions that cause serious disability without necessarily being life threatening: stroke closed head or spinal cord injuries mental retardation congenital malformations.

  o Conditions that cause significant pain or discomfort that can cause serious interruptions to life activities: severe allergies migraine arthritis sickle cell disease

  o Conditions that require major commitments of time and effort from care-givers for a substantial period of time: mobility disorders blindness Alzheimer's disease and other dementias chronic obstructive pulmonary disease paraplegia or quadriplegia Down's syndrome depression

  o Conditions that may require frequent monitoring: diabetes conditions requiring anticoagulation treatment severe asthma severe allergies schizophrenia and other psychotic illnesses.

  o Conditions that predict or are associated with severe consequences: hypertension (associated with heart disease) depression (associated with suicide) diabetes (associated with blindness, kidney failure) alcohol and other substance abuse (associated with intentional and unintentional injuries).
* Recent history of suspected substance abuse or a lifetime history of psychostimulant abuse and/or dependence
* Metal implants or braces (as determined through fMRI screening form)

Anorexia Nervosa

* Pregnancy or breast feeding within last 3 months
* Lifetime history of bipolar disorder or psychosis
* Illiterate/Blind individuals
* Contraindications to amisulpride or bromocriptine (as determined through medical history in bioscreen and PI interview) including: Syncopal migraine; Uncontrolled hypertension; Pheochromocytoma; Prolactinoma; Breast cancer; hypersensitivity/allergy to amisulpride or bromocriptine; History of long QT syndrome; Family history of sudden death or long QT syndrome; History of seizures or seizure disorder
* Use of an anti-psychotic or other dopamine acting medication including stimulants within the past week at time of MRI
* Recent history of substance abuse or dependence (within the last month)
* Major Medical illness (as determined through medical history in bioscreen and PI interview) such as:

  o Conditions that are life threatening: cancer heart disease stroke HIV/AIDS

  o Conditions that are life threatening Conditions that cause serious disability without necessarily being life threatening: stroke closed head or spinal cord injuries mental retardation congenital malformations.

  o Conditions that cause significant pain or discomfort that can cause serious interruptions to life activities: severe allergies migraine arthritis sickle cell disease

  o Conditions that require major commitments of time and effort from care-givers for a substantial period of time: mobility disorders blindness Alzheimer's disease and other dementias chronic obstructive pulmonary disease paraplegia or quadriplegia Down's syndrome

  o Conditions that may require frequent monitoring: diabetes conditions requiring anticoagulation treatment severe asthma severe allergies schizophrenia and other psychotic illnesses.

  o Conditions that predict or are associated with severe consequences: hypertension (associated with heart disease) diabetes (associated with blindness, kidney failure) alcohol and other substance abuse (associated with intentional and unintentional injuries) within the last month
* Metal implants or braces (as determined through fMRI screening form)

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 individuals were recruited and enrolled in the study between 10/20/2020 and 6/22/2023 from the San Diego community and the UC San Diego Health Eating Disorders Center for Treatment and Research. Subjects completed several screening processes to determine eligibility and after eligibility was confirmed, were randomly assigned to the study arms. Of those not randomized, 18 individuals were excluded (10 screen failures, 1 voluntary withdrawal by subject, and 7 withdrawals by PI).
Pre-assignment Details: Of the 31 subjects enrolled, 13 subjects were randomized, 7 participants in the healthy control group and 6 participants in the anorexia nervosa group. Each subject was assigned randomly to one of the 6 study arms. These study arms had different orders of the medication intervention administered at each scan. All subjects received each of the 3 study interventions (amysulpride, bromocriptine, placebo), however, the order of medication intervention at each scan varied based on the randomization.
Groups:
- Healthy Controls: Subjects at normal weight without psychiatric or eating disorder history
- Anorexia Nervosa: Subjects diagnosed with restricting-type anorexia nervosa according to DSM-V criteria
Period: 1st Intervention (1 Day)
Arm/Group | Healthy Controls | Anorexia Nervosa
Started | 7 | 6
1st Intervention = Amysulpride | 3 | 2
1st Intervention = Bromocriptine | 1 | 2
1st Intervention = Placebo | 3 | 2
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout Period (2-3 Days)
Arm/Group | Healthy Controls | Anorexia Nervosa
Started (There was a two to three day period in between each of the study scans in order to wash out the 1st intervention medication prior to the next scan intervention 2.) | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: 2nd Intervention (1 Day)
Arm/Group | Healthy Controls | Anorexia Nervosa
Started | 7 | 6
2nd Intervention = Amysulpride. | 2 | 2
2nd Intervention = Bromocriptine | 3 | 2
2nd Intervention = Placebo | 2 | 2
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout Period (2-3 Days)
Arm/Group | Healthy Controls | Anorexia Nervosa
Started (There was a two to three day period in between each of the study scans in order to wash out the 2nd intervention medication prior to the next scan and 3rd Intervention.) | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: 3rd Intervention (1 Day)
Arm/Group | Healthy Controls | Anorexia Nervosa
Started | 7 | 6
3rd Intervention = Amysulpride | 2 | 2
3rd Intervention = Bromocriptine | 3 | 2
3rd Intervention = Placebo | 2 | 2
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of baseline participants were the number of subjects who completed all the screening steps and were eligible for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Anorexia Nervosa | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.09 (4.02) | 21.43 (2.25) | 22.86 (3.47)
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were female in this study
  Participants
    Female | 7 | 6 | 13
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity Information
  Participants
    Hispanic or Latino | 3 | 2 | 5
    Not Hispanic or Latino | 4 | 4 | 8
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race information
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 4 | 4 | 8
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.41 (1.69) | 18.63 (0.94) | 20.67 (2.38)
Eating Disorder Inventory 3 - Drive for Thinness Subscale [Mean (Standard Deviation); unit: units on a scale] — The Eating Disorders Inventory (EDI-3) is a 91-question self-report measure that assesses the presence of eating disorders and eating disorder thoughts and behaviors. The drive for thinness subscale on the Eating Disorders Inventory 3 ranges from 0 to 28 with higher scores indicating worse outcome.
  units on a scale | 0.57 (0.79) | 19.5 (4.41) | 9.30 (10.24)
Eating Disorder Inventory 3 - Body Dissatisfaction Subscale [Mean (Standard Deviation); unit: units on a scale] — The Eating Disorders Inventory (EDI-3) is a 91-question self-report measure that assesses the presence of eating disorders and eating disorder thoughts and behaviors. The Body Dissatisfaction subscale on the Eating Disorders Inventory 3 ranges from 0 to 40 with higher scores indicating worse outcome.
  units on a scale | 5.00 (3.78) | 30.33 (4.76) | 16.69 (13.76)
Eating Disorders Examination Questionnaire Global Score [Mean (Standard Deviation); unit: units on a scale] — The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire, adapted from the semi-structured interview, the Eating Disorder Examination (EDE). The questionnaire is designed to assess the range, frequency and severity of behaviors associated with a diagnosis of an eating disorder. The overall global score ranges from 0 to 6 and is calculated by taking the average of all questions in the measure, with a higher score indicating more problematic eating difficulties.
  units on a scale | 0.33 (0.41) | 3.62 (0.88) | 1.85 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Brain Activation (Measured in Percent Signal Change) During a Prediction Error Taste Reward Task Using Functional Magnetic Resonance Imaging (fMRI).
Description: This task measures responsiveness to unexpected stimulus in the dopamine related brain circuitry. Study participants in both the healthy control group and anorexia nervosa group completed 3 fMRI scans. Prior to each scan subjects were administered one of three study medications (amisulpride, bromocriptine, or placebo). During the fMRI scan, subjects completed a taste reward prediction error task where they viewed visual stimuli and then received one of three conditions: sweet taste, neutral taste, or no solution. 20 percent of stimulus receipt was unexpected, that is there is a mismatch between expectation and outcome. Using a region of interest (ROI)-based approach, brain activation percent signal change values were extracted from the brain images for each subject and compared across groups and medication scans. A repeated measures ANOVA was used to calculate the mean brain activation for each group and each medication scan.
Time Frame: The outcome measure was assessed during the taste MRI task on each of the 3 intervention scan days over the course of 9 to 12 days
Population: brain imaging data was pre-processed and brain response was analyzed across groups (healthy control group versus anorexia nervosa group) and within group for each medication. One participant in the anorexia nervosa group had to be excluded from the analysis results due to excessive movement throughout the MRI scan.
Measure: Mean (Standard Error); unit: Percent Signal Change
Groups:
- Healthy Controls Placebo Scan: Subjects at normal weight without psychiatric or eating disorder history. Placebo medication was administered 3 hours prior to the start of the functional magnetic resonance imaging (fMRI) Taste Reward Task.
- Anorexia Nervosa Placebo Scan: Subjects diagnosed with restricting-type anorexia nervosa according to DSM-V criteria. Placebo medication was administered 3 hours prior to the start of the functional magnetic resonance imaging (fMRI) Taste Reward Task.
- Healthy Controls Amisulpride Medication Scan: Subjects at normal weight without psychiatric or eating disorder history. Amisulpride medication was administered 3 hours prior to the start of the functional magnetic resonance imaging (fMRI) Taste Reward Task.
- Anorexia Nervosa Amisulpride Medication Scan: Subjects diagnosed with restricting-type anorexia nervosa according to DSM-V criteria. Amisulpride medication was administered 3 hours prior to the start of the functional magnetic resonance imaging (fMRI) Taste Reward Task.
- Healthy Controls Bromocriptine Medication Scan: Subjects at normal weight without psychiatric or eating disorder history. Bromocriptine medication was administered 3 hours prior to the start of the functional magnetic resonance imaging (fMRI) Taste Reward Task.
- Anorexia Nervosa Bromocriptine Medication Scan: Subjects diagnosed with restricting-type anorexia nervosa according to DSM-V criteria. Bromocriptine medication was administered 3 hours prior to the start of the functional magnetic resonance imaging (fMRI) Taste Reward Task.
Arm/Group | Healthy Controls Placebo Scan | Anorexia Nervosa Placebo Scan | Healthy Controls Amisulpride Medication Scan | Anorexia Nervosa Amisulpride Medication Scan | Healthy Controls Bromocriptine Medication Scan | Anorexia Nervosa Bromocriptine Medication Scan
Number analyzed (Participants) | 7 | 5 | 7 | 5 | 7 | 5
Percent Signal Change
  Left Ventral Insula Brain Activation | 5.847 (1.349) | 5.083 (1.596) | 0.991 (0.938) | -1.047 (1.109) | 1.116 (1.225) | -0.148 (1.450)
  Right Ventral Insula Brain Activation | 4.095 (0.669) | 4.860 (0.791) | 0.883 (0.716) | -0.137 (0.847) | 4.117 (0.987) | 2.650 (1.167)
  Left Ventral Striatum Brain Activation | 2.081 (0.582) | 1.767 (0.689) | 1.475 (1.153) | -0.599 (1.365) | 1.122 (0.951) | 1.328 (1.126)
  Right Ventral Striatum Brain Activation | 1.583 (0.660) | 2.367 (0.781) | 1.728 (1.020) | -0.799 (1.207) | 1.642 (0.304) | 1.732 (0.359)
  Left Inferior Orbital Frontal Cortex Brain Activation | -0.199 (0.789) | 0.544 (0.934) | 0.988 (0.686) | -1.222 (0.811) | 0.646 (1.038) | 1.171 (1.229)
  Right Inferior Orbital Frontal Cortex Brain Activation | 4.333 (0.427) | 4.138 (0.505) | 0.396 (0.803) | -0.699 (0.950) | 5.512 (1.244) | 4.774 (1.472)

2. Primary Outcome: Measurement of Brain Activation (Measured in Percent Signal Change) During Taste Stimulus Expectation Using Functional Magnetic Resonance Imaging (fMRI).
Description: Study participants in both the healthy control group and anorexia nervosa group completed 3 fMRI scans. Prior to each scan subjects were administered one of three study medications (amisulpride, bromocriptine, or placebo). During the fMRI scan, subjects completed a taste reward prediction error task where they viewed visual stimuli and then received one of three conditions: sweet taste, neutral taste, or no solution. Using a region of interest (ROI)-based approach, brain activation percent signal change values were extracted from the brain images for each subject and compared across groups and medication scans. Here only stimulus expectation data were analyzed. A repeated measures ANOVA was used to calculate the mean brain activation for each group and each medication scan.
Time Frame: as for outcome 1
Population: brain imaging data was pre-processed and brain response was analyzed across groups (healthy control group versus anorexia nervosa group) and within group for each medication
Measure: Mean (Standard Error); unit: Percent Signal Change
Arm/Group | Healthy Controls Placebo Scan | Anorexia Nervosa Placebo Scan | Healthy Controls Bromocriptine Medication Scan | Anorexia Nervosa Bromocriptine Medication Scan | Healthy Controls Amisulpride Medication Scan | Anorexia Nervosa Amisulpride Medication Scan
Number analyzed (Participants) | 7 | 5 | 7 | 5 | 7 | 5
Percent Signal Change
  Left Ventral Insula Brain Activation | 4.799 (0.681) | 3.282 (0.806) | 4.821 (1.481) | 5.569 (1.752) | 5.265 (0.803) | 4.691 (0.950)
  Right Ventral Insula Brain Activation | 3.884 (0.526) | 3.015 (0.622) | 4.436 (2.406) | 5.866 (2.847) | 3.464 (0.725) | 3.383 (0.858)
  Left Ventral Striatum Brain Activation | 1.558 (0.347) | 1.790 (0.411) | 3.450 (1.174) | 2.860 (1.390) | 1.206 (0.390) | 1.738 (0.461)
  Right Ventral Striatum Brain Activation | 1.717 (0.381) | 1.501 (0.451) | 4.700 (1.459) | 3.208 (1.727) | 2.163 (0.758) | 1.609 (0.897)
  Left Inferior Orbital Frontal Cortex Brain Activation | 3.649 (0.480) | 2.259 (0.569) | 3.838 (2.061) | 6.392 (2.439) | 3.562 (0.996) | 4.722 (1.178)
  Right Inferior Orbital Frontal Cortex Brain Activation | 4.193 (0.782) | 3.352 (0.926) | 4.745 (1.758) | 5.712 (2.080) | 5.362 (1.130) | 4.226 (1.337)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed from the administration of the medication on scan 1 (1st intervention) through the end of scan 3 (3rd intervention). The time period was 9 to 12 days depending on length of each washout period.
Groups:
- Healthy Control Group Placebo Scan: Healthy Control subjects were administered placebo 3 hours prior to the start of the MRI. Subjects performed prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
- Anorexia Nervosa Group Placebo Scan: Anorexia Nervosa subjects were administered placebo pill 3 hours prior to the start of the MRI. Subjects performed prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
- Healthy Control Group Amisulpride Scan: Healthy Control subjects were administered the dopamine D2 antagonist medication amisulpride 3 hours prior to the start of the MRI. Subjects performed prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
- Anorexia Nervosa Group Amisulpride Scan: Anorexia Nervosa subjects were administered the dopamine D2 antagonist medication amisulpride 3 hours prior to the start of the MRI. Subjects performed prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
- Healthy Control Group Bromocriptine Scan: Healthy Control subjects were administered the dopamine D2 receptor agonist medication bromocriptine 3 hours prior to the start of the MRI. Subjects performed prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
- Anorexia Nervosa Group Bromocriptine Scan: Anorexia Nervosa subjects were administered the dopamine D2 receptor agonist medication bromocriptine 3 hours prior to the start of the MRI. Subjects performed prediction error and reversal tasks during functional magnetic resonance imaging (fMRI).
Arm/Group | Healthy Control Group Placebo Scan | Anorexia Nervosa Group Placebo Scan | Healthy Control Group Amisulpride Scan | Anorexia Nervosa Group Amisulpride Scan | Healthy Control Group Bromocriptine Scan | Anorexia Nervosa Group Bromocriptine Scan
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/6 | 2/7 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control Group Placebo Scan (N=7) | Anorexia Nervosa Group Placebo Scan (N=6) | Healthy Control Group Amisulpride Scan (N=7) | Anorexia Nervosa Group Amisulpride Scan (N=6) | Healthy Control Group Bromocriptine Scan (N=7) | Anorexia Nervosa Group Bromocriptine Scan (N=6)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT04128683/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT04128683/ICF_001.pdf